CLINICAL TRIAL: NCT05735002
Title: PRomoting Early Diagnosis Of Chronic Mesenteric ISchEmia by a Mesenteric Artery Calcium Score Based Risk Stratification and Detection of Postprandial Mucosal Ischemia by Butyrate Breath Testing
Brief Title: Promoting Early Diagnosis of Chronic Mesenteric Ischemia
Acronym: PROMISE
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maag Lever Darm Stichting (Other)
Responsible Party: Principal Investigator, Marco J. Bruno, Gastroenterologist, Erasmus Medical Center
Other Study IDs: 9933
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Chronic Mesenteric Ischemia
Keywords: breath test, chronic mesenteric ischemie, calcium scoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected to search for specific biomarkers for chronic mesenteric ischemia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected CMI: Patients with suspected CMI
  Interventions: Diagnostic Test: 13C-butyrate breath test

INTERVENTIONS:
Diagnostic Test: 13C-butyrate breath test — breath test

SUMMARY:
CMI is an incapacitating disease and timely diagnosis remains problematic. Despite the substantial compensatory capacity of the mesenteric circulation CMI is relatively common, its incidence being comparable to other well-known diseases like Crohn's disease.

Diagnostic tools are needed for two purposes since the exclusion of CMI currently requires a cumbersome complication-prone diagnostic workup and since a definitive diagnosis is mainly established per exclusionem. First, a sensitive test is desirable to rule out CMI and avoid excessive diagnostic investigations. Quantification of mesenteric arterial calcification on computed tomography (CT) seems suitable for this purpose, synonymous with the coronary artery calcium score. Second, a specific test is required confirming CMI by detection of mucosal ischemia during a meal, when oxygen demand peaks. A breath test, based on the requirement of oxygen to absorb and metabolize 13C-butyrate in the enterocyte, could detect mucosal ischemia

Objective: Facilitating diagnosis of chronic mesenteric ischemia (CMI) using 1) the mesenteric artery calcium score (MACS) and 2) mucosal ischemia detection by butyrate breath testing

Study design: Multicentre prospective cohort studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical suspicion of CMI referred to Maagdarm Ischemie Centrum Rotterdam (MICR), MST or UMCG.
* Patients ≥ 18 years

Exclusion Criteria:

* Patients who are unable to give informed consent
* Patients with previous mesenteric artery revascularization
* No available CT imaging and contraindications for CT imaging (e.g. pregnancy)
* Common origin of the celiac artery and superior mesenteric artery
* Known delayed gastric emptying
* Known and untreated small intestinal bacterial overgrowth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspected CMI
Sampling Method: Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Breath test | 2023-2025
  - To validate the butyrate breath test as a specific functional test with a high positive predictive value to rightfully diagnose and select patients who will benefit from invasive treatment.
calcium scores | 2023-2035
  To validate the mesenteric artery calcium score as a readily available, easy, and sensitive test with a high negative predictive value to either rule out CMI or select patients for further investigations.

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Medisch Spectrum Twente, Enschede, Overijssel
  - University Medical Centre Groningen, Groningen, Provincie Groningen
  - Erasmus University Medical Centre Rotterdam, Rotterdam, South Holland
  - Franciscus, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided